CLINICAL TRIAL: NCT02349061
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Proof-of-Concept Study of Ustekinumab in Subjects With Active Systemic Lupus Erythematosus
Brief Title: A Phase 2a, Efficacy and Safety Study of Ustekinumab in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR106661; CNTO1275SLE2001 (Other: Janssen Research & Development, LLC); 2014-005000-19 (EudraCT Number)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus; Ustekinumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Ustekinumab plus Concomitant Medication (Experimental): Participants will receive weight-range based dosing of approximately 6 mg/kg of ustekinumab intravenously at Week 0 followed by ustekinumab 90 mg subcutaneously (SC) every 8 weeks (q8w) up to Week 40. Participants who meet the study extension inclusion criteria will continue to receive ustekinumab 90 mg SC q8w starting at Week 48 or 56 through Week 104. Participants will continue stable concomitant treatment through Week 48, as well as through the study extension although tapering of corticosteroids is encouraged beyond Week 48. Participants who complete or discontinue study treatment will be evaluated for 16 additional Weeks of safety follow-up.
  Interventions: Drug: Ustekinumab IV; Drug: Ustekinumab SC; Other: Concomitant Medication
- Placebo followed by Ustekinumab plus Concomitant Medication (Experimental): Participants will receive placebo intravenously at Week 0 followed by placebo subcutaneously at Weeks 8 and 16. At week 24 participants will receive ustekinumab SC q8w up to Week 40. Participants who meet the study extension inclusion criteria will continue to receive ustekinumab 90 mg SC q8w starting at Week 48 or 56 through Week 104. Participants will continue stable concomitant treatment through Week 48, as well as through the study extension although tapering of corticosteroids is encouraged beyond Week 48. Participants who complete or discontinue study treatment will be evaluated for 16 additional Weeks of safety follow-up.
  Interventions: Drug: Placebo Infusion; Drug: Placebo SC; Drug: Ustekinumab SC; Other: Concomitant Medication

INTERVENTIONS:
Drug: Ustekinumab IV — Weight-range based dosing of approximately 6 mg/kg of ustekinumab intravenously at Week 0.
  Other Names: STELARA
  Arms: Ustekinumab plus Concomitant Medication
Drug: Placebo Infusion — Placebo intravenously at Week 0.
  Arms: Placebo followed by Ustekinumab plus Concomitant Medication
Drug: Placebo SC — Placebo subcutaneously at Weeks 8 and 16.
  Arms: Placebo followed by Ustekinumab plus Concomitant Medication
Drug: Ustekinumab SC — Ustekinumab 90 mg subcutaneously every 8 weeks up to Week 40 and up to Week 104 in study extension (for eligible participants)
Other: Concomitant Medication — Concomitant treatment (mycophenolate, azathioprine/6-mercaptopurine, methotrexate, hydroxychloroquine and/or chloroquine, oral corticosteroids, NSAIDs, antihypertensive medications, and topical medications) through Week 48, as well as through the study extension although tapering of corticosteroids is encouraged beyond Week 48.

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab as measured by a reduction in disease activity for subjects with active Active Systemic Lupus Erythematosus (SLE - chronic disorder of connective tissue in which there can be skin rash, arthritis, kidney problems, and anemia, among other problems).

DETAILED DESCRIPTION:
A multicenter (more than one medical research center involved in study), randomized (study drug assigned by chance), double-blind (neither the Investigator nor the participant know about the study drug), placebo-controlled, proof-of-concept study of ustekinumab in participants with active systemic lupus erythematosus. Participants will be screened to achieve all inclusion criteria and none exclusion criteria and will then receive either ustekinumab or placebo along with concomitant background medicine. Participants will be primarily assessed for response using the Systemic Lupus Erythematosus Response Index 2000 (SRI-4). Participants' safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented medical history to meet SLICC classification criteria for SLE for a minimum of 3 months prior to first dose
* At least 1 well-documented (subject file, referring physician letter, or laboratory result), unequivocally positive, documented test for autoantibodies in medical history including either of the following: ANA, and/or anti-dsDNA antibodies, and/or anti-Smith antibodies
* At least 1 unequivocally positive autoantibody test including ANA and/or anti-dsDNA antibodies and/or anti-Smith antibodies detected during screening
* At least 1 BILAG A and/or 2 BILAG B domain scores observed during screening prior to first administration of study agent
* Demonstrate active disease based on SLEDAI-2K score greater than or equal to (>=) 6 observed during screening and assessed approximately 2 to 6 weeks prior to randomization. Must also have SLEDAI-2K score >= 4 for clinical features (ie, SLEDAI excluding laboratory results) at Week 0 prior to the first administration of study agent

Exclusion Criteria:

* Have other inflammatory diseases that might confound the evaluations of efficacy, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis (PsA), RA/lupus overlap, psoriasis or active Lyme disease
* Are pregnant, nursing, or planning a pregnancy or fathering a child while enrolled in the study or within 4 months after receiving the last administration of study agent
* Have received systemic or topical cream/ointment preparations of cyclosporine A or other systemic immunomodulatory agents other than those described in inclusion criteria within the past 3 months prior to first administration of study agent
* Have received a single B cell targeting agent within 3 months prior to first study agent administration; or received more than 1 previous B cell targeting therapy including belimumab or epratuzamab within 6 months prior to first administration of the study agent; or received B cell depleting therapy (eg, rituximab) within 12 months prior to first administration of the study agent or have evidence of continued B-cell depletion following such therapy
* Have ever received ustekinumab
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin that has been treated with no evidence of recurrence for at least 3 months before the first study agent administration and carcinoma in situ of the cervix that has been surgically cured)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (43):
- United States (12):
  - Huntsville, Alabama
  - Beverly Hills, California
  - Tampa, Florida
  - Lansing, Michigan
  - Manhasset, New York
  - New York, New York
  - Syracuse, New York
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Jackson, Tennessee
- Argentina (3):
  - Buenos Aires
  - Ciudad de San Miguel de Tucuman
  - San Juan
- Australia (5):
  - Adelaide
  - Camberwell
  - Heidelberg
  - Liverpool
  - Nedlands
- Germany (3):
  - Berlin
  - Cologne
  - Frankfurt
- Hungary (4):
  - Budapest
  - Debrecen
  - Szeged
  - Zalaegerszeg
- Mexico (4):
  - Chihuahua City
  - Guadalajara
  - León
  - México
- Poland (4):
  - Bydgoszcz
  - Poznan
  - Szczecin
  - Wroclaw
- Spain (5):
  - Barcelona
  - Madrid
  - Málaga
  - Santiago de Compostela
  - Seville
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taoyuan District

REFERENCES:
- [Derived] van Vollenhoven RF, Hahn BH, Tsokos GC, Lipsky P, Gordon RM, Fei K, Lo KH, Chevrier M, Rose S, Berry P, Yao Z, Karyekar CS, Zuraw Q. Efficacy and Safety of Ustekinumab in Patients With Active Systemic Lupus Erythematosus: Results of a Phase II Open-label Extension Study. J Rheumatol. 2022 Apr;49(4):380-387. doi: 10.3899/jrheum.210805. Epub 2021 Dec 1. PMID 34853089
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Cesaroni M, Seridi L, Loza MJ, Schreiter J, Sweet K, Franks C, Ma K, Orillion A, Campbell K, M Gordon R, Branigan P, Lipsky P, van Vollenhoven R, Hahn BH, Tsokos GC, Chevrier M, Rose S, Baribaud F, Jordan J. Suppression of Serum Interferon-gamma Levels as a Potential Measure of Response to Ustekinumab Treatment in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2021 Mar;73(3):472-477. doi: 10.1002/art.41547. Epub 2021 Feb 1. PMID 33010188
- [Derived] van Vollenhoven RF, Hahn BH, Tsokos GC, Lipsky P, Fei K, Gordon RM, Gregan I, Lo KH, Chevrier M, Rose S. Maintenance of Efficacy and Safety of Ustekinumab Through One Year in a Phase II Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled Crossover Trial of Patients With Active Systemic Lupus Erythematosus. Arthritis Rheumatol. 2020 May;72(5):761-768. doi: 10.1002/art.41179. Epub 2020 Apr 1. PMID 31769212
- [Derived] van Vollenhoven RF, Hahn BH, Tsokos GC, Wagner CL, Lipsky P, Touma Z, Werth VP, Gordon RM, Zhou B, Hsu B, Chevrier M, Triebel M, Jordan JL, Rose S. Efficacy and safety of ustekinumab, an IL-12 and IL-23 inhibitor, in patients with active systemic lupus erythematosus: results of a multicentre, double-blind, phase 2, randomised, controlled study. Lancet. 2018 Oct 13;392(10155):1330-1339. doi: 10.1016/S0140-6736(18)32167-6. Epub 2018 Sep 21. PMID 30249507

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 participants were screened during the study, 102 were enrolled/randomized and treated.
Groups:
- Placebo - Ustekinumab: Participants received placebo matched to ustekinumab intravenously (IV) at Week 0 then followed by placebo subcutaneously (SC) at Week 8 and 16. At Week 24, participants who completed were crossed-over to receive ustekinumab 90 milligram (mg) SC at Weeks 24, 32, and 40 followed by safety follow-up through Week 56 in a blinded fashion for 16 weeks after last study agent SC administration.
- Ustekinumab: Participants received an initial body weight range based IV dose approximating 6 milligram per kilogram (mg/kg) of ustekinumab at Week 0 followed by 90 mg SC administered every 8 weeks (q8w) at Weeks 8 and 16. Participants who completed placebo controlled period (PCP) continued to receive ustekinumab 90 mg at Weeks 24, 32, and 40 followed by safety follow-up for 16 weeks after last study agent SC administration. Per the amended study design, open-label ustekinumab 90 mg q8w SC administration will continue to be provided through Week 104 (study extension) to eligible participants followed by safety follow-up through Week 120.
- Placebo to Ustekinumab: Participants who received placebo matched to ustekinumab and completed PCP period in placebo group were crossed-over at Week 24 and received ustekinumab 90 mg SC at Weeks 24, 32, and 40 followed by safety follow-up through Week 56 in a blinded fashion for 16 weeks after last study agent SC administration. Per the amended study design, open-label ustekinumab 90 mg q8w SC administration will continue to be provided through Week 104 (study extension) to eligible participants followed by safety follow-up through Week 120.
Period: Main Study: PCP (Up to Week 24)
Arm/Group | Placebo - Ustekinumab | Ustekinumab | Placebo to Ustekinumab
Started | 42 | 60 | 0
Completed | 33 | 56 | 0
Not Completed | 9 | 4 | 0
Not completed — Adverse Event | 4 | 3 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Main Study: Week 24 to 56
Arm/Group | Placebo - Ustekinumab | Ustekinumab | Placebo to Ustekinumab
Started | 0 | 56 | 33
Completed | 0 | 53 | 30
Not Completed | 0 | 3 | 3
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Period: Study Extension (Week 56 to Week 120)
Arm/Group | Placebo - Ustekinumab | Ustekinumab | Placebo to Ustekinumab
Started | 0 | 29 (Who met study extension inclusion criteria received open-label ustekinumab SC through Week 104.) | 17 (Who met study extension inclusion criteria received open-label ustekinumab SC through Week 104.)
Completed | 0 | 24 | 14
Not Completed | 0 | 5 | 3
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Ustekinumab | Ustekinumab | Total
Number analyzed (Participants) | 42 | 60 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.03) | 40 (11.95) | 41.3 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 58 | 93
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 20 | 32
  Not Hispanic or Latino | 30 | 40 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 28 | 42 | 70
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 8 | 14
  Black or African American | 3 | 4 | 7
  Hispanic or Latino | 7 | 13 | 20
  Other | 5 | 6 | 11
  White Non-Hispanic | 21 | 29 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 4 | 8 | 12
  Australia | 2 | 3 | 5
  Germany | 2 | 3 | 5
  Hungary | 4 | 4 | 8
  Mexico | 6 | 5 | 11
  Poland | 7 | 12 | 19
  Spain | 5 | 7 | 12
  Taiwan, Province Of China | 6 | 7 | 13
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Systemic Lupus Erythematosus Responder Index (SRI-4) Composite Response (CR) at Week 24
Description: SRI-4 response was defined as greater than or equal to 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score and no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA). Composite response is defined as SRI-4 response in participants who do not meet treatment failure criteria. SLEDAI-2K assessment consists of 24 items with total score of 0 to 105, with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale = from very well (0)-very poor (10).
Time Frame: Week 24
Population: Full analysis set (FAS) included all the randomized participants who received at least 1 dose (partial or complete, IV or SC) of ustekinumab or placebo.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants received placebo matched to ustekinumab intravenously (IV) at Week 0 then followed by placebo subcutaneously (SC) at Week 8 and 16.
- Ustekinumab: Participants received an initial body weight range based IV dose approximating 6 milligram per kilogram (mg/kg) of ustekinumab at Week 0 followed by 90 mg SC administered every 8 weeks (q8w) at Weeks 8 and 16.
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 42 | 60
Percentage of participants | 33.3 | 61.7
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab; Test type: Superiority; p = 0.0057, Regression, Logistic; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.41 to 7.63]

2. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K) Score at Week 24
Description: The SLEDAI-2K is an established, validated SLE activity index. It is based on the presence of 24 features in 9 organ systems and measures disease activity in SLE patients in the previous 30 days. It is weighted according to the feature. Features are scored by the assessing physician if present within the last 30 days with more severe features having higher scores, and then simply added to determine the total SLEDAI 2K score, which ranges from 0 to 105, with higher scores representing increased disease activity.
Time Frame: Baseline, Week 24
Population: FAS included all the randomized participants who received at least 1 dose (partial or complete, IV or SC) of ustekinumab or placebo. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 31 | 53
Units on a scale | -3.8 (5.39) | -4.4 (2.91)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab; Test type: Superiority; p = 0.0929, Mixed model repeated measures model; Least Squares (LS) Mean Difference = -1.36, 95% CI 2-sided [-2.94 to 0.23]

3. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (PGA) Score at Week 24
Description: PGA was recorded on a visual analogue scale (VAS; 0.0 to 10.0 centimeter [cm]). The scale for the physician's assessment ranges for 'no lupus activity' (0.0) to 'extremely active lupus' (10.0).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 32 | 55
Units on a scale | -1.93 (2.168) | -2.17 (1.915)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab; Test type: Superiority; p = 0.3944, Mixed model repeated measures model; LS Means Difference = -0.383, 95% CI 2-sided [-1.271 to 0.506]

4. Secondary Outcome: Number of Participants With BILAG-based Combined Lupus Assessment (BICLA) Response at Week 24
Description: BICLA response defined as participants meeting following criteria: 1. BILAG improvement (all BILAG A scores at baseline improved to either B, C or D and all BILAG B scores at baseline improved to C or D and no worsening in disease activity defined as no new BILAG A scores and <= 1 new BILAG B score) and 2. no worsening of total SLEDAI-2K from baseline 3. < 1 cm increase in PGA and 4. no treatment failure criteria met. BILAG: assesses disease extent, severity (range: A [severe] to E [no disease]). SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). PGA: assesses worsening in participant's general health status (0.0= 'no lupus activity' to 10.0 = 'extremely active lupus').
Time Frame: Week 24
Population: FAS included all the randomized participants who received at least 1 dose (partial or complete, IV or SC) of ustekinumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 42 | 60
Participants | 14 | 21
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab; Test type: Superiority; p = 0.9939, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.43 to 2.34]

5. Secondary Outcome: Change From Baseline in Number of Joints With Pain and Signs of Inflammation at Week 24
Description: Change from baseline in number of joints (active joint) with pain and signs of inflammation (tenderness, swelling or effusion) for participants with at least 2 affected joints at baseline were reported. An active joint is defined as a joint with pain and signs of inflammation (e.g., tenderness, swelling or effusion).
Time Frame: Baseline, Week 24
Population: FAS included all the randomized participants who received at least 1 dose (partial or complete, IV or SC) of ustekinumab or placebo. Population included participants with at least 2 affected joints at baseline (2 or more affected joints).
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo | Ustekinumab
Number analyzed (Participants) | 31 | 51
Joints | -2.8 (7.31) | -4.5 (4.42)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab; Test type: Superiority; p = 0.1032, Mixed model repeated measures model; LS Means Difference = -2.17, 95% CI 2-sided [-4.78 to 0.45]

ADVERSE EVENTS:
Time Frame: Screening up to Week 120
Description: Safety analysis set was defined as the set of all randomized participants who have received at least 1 dose (partial or complete, intravenously [IV] or subcutaneously [SC]) of ustekinumab or placebo.
Groups:
- Placebo (Up to Week 24): Participants received placebo matched to ustekinumab intravenously (IV) at Week 0 then followed by placebo subcutaneously (SC) at Week 8 and 16.
- Ustekinumab (Up to Week 24): Participants received an initial body weight range based IV dose approximating 6 milligram per kilogram (mg/kg) of ustekinumab at Week 0 followed by 90 mg SC administered every 8 weeks (q8w) at Week 8 and 16.
- Placebo to Ustekinumab (Week 24 to 56): Participants who received placebo matched to ustekinumab and completed placebo controlled period (PCP) in placebo group were crossed-over at Week 24 and received ustekinumab 90 milligram (mg) SC at Weeks 24, 32, and 40 followed by safety follow-up through Week 56 in a blinded fashion for 16 weeks after last study agent SC administration.
- Ustekinumab (Week 24 to 56): Participants who were assigned to Ustekinumab treatment and who completed PCP continued to receive ustekinumab 90 mg SC at Weeks 24, 32, and 40 followed by safety follow up for 16 weeks after last study agent SC administration.
- Placebo to Ustekinumab (Week 56 to 120); Ustekinumab (Week 56 to 120): Per the amended study design, open-label ustekinumab 90 mg q8w SC administration will continue to be provided through Week 104 (study extension) to eligible participants followed by safety follow-up through Week 120.
Arm/Group | Placebo (Up to Week 24) | Ustekinumab (Up to Week 24) | Placebo to Ustekinumab (Week 24 to 56) | Ustekinumab (Week 24 to 56) | Placebo to Ustekinumab (Week 56 to 120) | Ustekinumab (Week 56 to 120)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/60 | 0/33 | 0/56 | 0/17 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/42 | 5/60 | 5/33 | 7/56 | 1/17 | 4/29
Other Adverse Events (participants affected / at risk) | 25/42 | 30/60 | 21/33 | 34/56 | 8/17 | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to Week 24) (N=42) | Ustekinumab (Up to Week 24) (N=60) | Placebo to Ustekinumab (Week 24 to 56) (N=33) | Ustekinumab (Week 24 to 56) (N=56) | Placebo to Ustekinumab (Week 56 to 120) (N=17) | Ustekinumab (Week 56 to 120) (N=29)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Salmonella Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Stenotrophomonas Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lupus Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Raynaud's Phenomenon (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to Week 24) (N=42) | Ustekinumab (Up to Week 24) (N=60) | Placebo to Ustekinumab (Week 24 to 56) (N=33) | Ustekinumab (Week 24 to 56) (N=56) | Placebo to Ustekinumab (Week 56 to 120) (N=17) | Ustekinumab (Week 56 to 120) (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 4 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 3 | 1 | 3
Dry Eye (Eye disorders) | 0 | 0 | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 1 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 4 | 0 | 4
Gastroenteritis (Infections and infestations) | 2 | 1 | 3 | 0 | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Infected Bite (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 2 | 6 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 3 | 1 | 1 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Tinea Versicolour (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 3
Tooth Infection (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 5 | 3 | 10 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 4 | 6 | 6 | 10 | 2 | 6
Vulvitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 1 | 1 | 2 | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 5 | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 1 | 2
Headache (Nervous system disorders) | 5 | 4 | 1 | 3 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 2
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication o r presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT02349061/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02349061/SAP_001.pdf